CLINICAL TRIAL: NCT02822157
Title: Circulating Tumor DNA Guiding (Olaparib) Lynparza® Treatment in Ovarian
Brief Title: Circulating Tumor DNA Guiding (Olaparib) Lynparza® Treatment in Ovarian Cancer
Acronym: CLIO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLIO
Record Dates: First submitted 2016-06-06; First posted 2016-07-04 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Ovarian Epithelial Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — olaparib; Carboplatin; Gemcitabine; Paclitaxel; liposomal doxorubicin; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olaparib (Experimental): olaparib 300mg oral tablets twice daily for 28 days in 28-day cycles
  Interventions: Drug: Olaparib
- Chemotherapy (Active Comparator): physician's choice chemotherapy
  Interventions: Drug: carboplatin + gemcitabine or carboplatin + paclitaxel or carboplatin + liposomal doxorubicin or liposomal doxorubicin 4-weekly or topotecan or paclitaxel weekly

INTERVENTIONS:
Drug: Olaparib
  Other Names: Lynparza
  Arms: Olaparib
Drug: carboplatin + gemcitabine or carboplatin + paclitaxel or carboplatin + liposomal doxorubicin or liposomal doxorubicin 4-weekly or topotecan or paclitaxel weekly — physician's choice chemotherapy
  Arms: Chemotherapy

SUMMARY:
This is a randomized, open-label, two-arm study in patients with relapsed epithelial ovarian tumors. Patients will be randomized in a 1:1 ratio to receive olaparib or standard chemotherapy with the possibility of crossover at the time of progression.

ELIGIBILITY:
Inclusion Criteria:

* with recurrent epithelial carcinoma of the ovary, fallopian tube or primary peritoneum
* At least 1 previous line of chemotherapy
* Measurable disease
* Patients have a normal organ and bone marrow function measured within 28 days of randomization
* WHO 0-2

Exclusion Criteria:

* Primary platinum-refractory disease
* Known hypersensitivity to olaparib
* Resting ECG with QTc > 470 msec
* Concomitant use of known potent CYP3A4 inhibitors
* Symptomatic uncontrolled brain metastases
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-08; Primary Completion 2021-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Overall Objective Response | 1 year after end inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Ignace Vergote, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZLeuven, Leuven, Belgium

REFERENCES:
- [Derived] Tattersall A, Ryan N, Wiggans AJ, Rogozinska E, Morrison J. Poly(ADP-ribose) polymerase (PARP) inhibitors for the treatment of ovarian cancer. Cochrane Database Syst Rev. 2022 Feb 16;2(2):CD007929. doi: 10.1002/14651858.CD007929.pub4. PMID 35170751